CLINICAL TRIAL: NCT03631680
Title: The Role of Estrogen in Adipocyte Remodeling Following Surgical Menopause
Acronym: RESUME
Status: Terminated | Type: Observational
Why Stopped: PI left the institution and the study was closed.
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana Clinical and Translational Science Center (Other)
Responsible Party: Principal Investigator, Kara Marlatt, Postdoctoral Researcher, Pennington Biomedical Research Center
Other Study IDs: PBRC 2018-022
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Menopause Surgical; Estrogen Deficiency; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 'Bilateral Oophorectomy Surgery' Group: Premenopausal women planning to undergo a laparoscopic, elective bilateral oophorectomy surgery.
  Interventions: Procedure: Bilateral Oophorectomy Surgery
- 'Comparative (Control)' Group: Premenopausal women with normal menstrual cycles from a previously completed study at Pennington Biomedical Research Center [NCT01748994] will serve as a comparator (control) group.

INTERVENTIONS:
Procedure: Bilateral Oophorectomy Surgery — Women undergoing elective, laparoscopic bilateral oophorectomy surgery will be enrolled.
  Groups: 'Bilateral Oophorectomy Surgery' Group

SUMMARY:
The overarching aim of this study is to assess the downstream effects of abrupt estrogen deficiency in women undergoing elective bilateral oophorectomy by studying:

1. the rate of in vivo adipogenesis in the subcutaneous abdominal (scABD) and subcutaneous femoral (scFEM) adipose tissue depots following bilateral oophorectomy surgery using an innovative (and tested) 8-week incorporation of stable isotope (deuterium; 2H) administered in the form of heavy water (2H2O) to endogenously label adipose tissue DNA;
2. the changes in expression of subcutaneous adipose tissue genes and proteins specific to adipocyte expansion and function; extracellular matrix remodeling and fibrosis; and inflammation in the scABD and scFEM depots before and after elective bilateral oophorectomy.

DETAILED DESCRIPTION:
This is a cross-sectional study that will enroll up to 10 women undergoing laparoscopic, elective bilateral oophorectomy at a local hospital in Baton Rouge, LA. Women will complete 7 study visits over 3 months; a single screening visit to assess eligibility, a pre-bilateral oophorectomy visit for imaging and adipose tissue biopsy collection, and 5 post-bilateral oophorectomy visits to "dose", maintain compliance and subject retention, and perform follow-up imaging and adipose tissue biopsy collection for outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females
* Ages 18-45 y
* BMI between 25 kg/m2 and 40 kg/m2 (±0.5 kg/m2 will be accepted)
* Are pre-menopausal (follicle-stimulating hormone, FSH<40 mIU/mL)
* Asymptomatic for the following menopause-related symptoms: hot flashes, insomnia (trouble sleeping), or mood swings
* Planning to have a laparoscopically, elective bilateral oophorectomy
* No medical indication for increased cancer risk
* Are willing to drink heavy water (2H2O) over an 8-week period
* Medically cleared for participation in the study by OB/GYN and Medical Investigator
* Are willing to have blood and fat tissue stored for future use

Exclusion Criteria:

* Unstable weight in the last 3 months [gain or loss >7 lb (or 3.2 kg)]
* Significant changes in diet or physical activity level within the past month
* Smoking or use of tobacco products within the last 3 months
* Amenorrhea (or absence of regular monthly cycles)
* History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
* Average screening blood pressure >140/90 mmHg
* Chronic use of systemic glucocorticoids, systemic adrenergic-stimulating agents, antipsychotic/antidepressant medications, thiazolidinediones, and other medications that cause clinically significant weight gain, weight loss or are known to make changes in fat cell number/size.
* Previous bariatric surgery (or other surgeries) for obesity or weight loss
* Use of over the counter or prescription weight loss products
* History of metabolic diseases (other than diabetes)
* History of neurological disease
* History of cardiovascular disease (or other chronic diseases)
* Unable or unwilling to have an MRI performed
* Pregnant, planning to become pregnant, or breastfeeding
* Use of hormone replacement therapy.
* Unwilling to discontinue any form or hormonal therapy (e.g., contraceptives including birth control pills, vaginal ring, injections, implant, or skin patch; hormonal supplements, etc.) upon enrollment (after the Screening Visit).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal women planning to undergo elective, laparoscopic bilateral oophorectomy surgery.
Study Population: Healthy women that are planning to undergo elective, laparoscopic bilateral oophorectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Rate of in vivo adipogenesis (via deuterium-enrichment of adipose tissue DNA) | Change from baseline in enrichment of DNA of adipose cells with deuterium at 8 weeks post-surgery
  Deuterium from the deuterium-labeled water is incorporated into the newly-synthesized DNA of newly-formed fat cell precursor cells through cell replication. The latter carry over the label when they become fat cells through differentiation. Enzymatic digestion of the fat tissue isolates the individual cells constituting the fat tissue. Centrifugation of the cell suspension allows the separation of fat cells into a floating layer and a pellet comprised of stromal-vascular cells including the fat cell precursor cells and small fat cells. As the fat cell precursor cells and small adipocytes have the property to attach quickly to plastic surfaces of culture dishes, a brief culturing of the stromal-vascular cells sorts these cells from the remaining cells. Thus, measuring the deuterium-enrichment of DNA from plastic-adherent stromal-vascular cells indicates the rate of in vivo formation of new mature fat cells and pre-adipocytes, a process collectively termed adipogenesis.

SECONDARY OUTCOMES:
Size of adipocytes | Change from baseline in size of adipocytes at 8 weeks post-surgery
  Fat cell size will be determined using osmium fixation of the lipids and measurement of their diameter with Coulter Counter followed by calculation of fat cell volume. The mean lipid content of fat cells will be calculated by multiplying the fat cell volume by the density of triolein (0.915).
Number of adipocytes | Change from baseline in number of adipocytes at 8 weeks post-surgery
  Fat cell number will be estimated by dividing the volume of adipose tissue depot of interest to the mean fat cell volume or the fat mass of the depot to the mean lipid content in fat cell.
Body composition (by Dual-energy X-ray Absorptiometry (DXA)) | Change from baseline in body composition at 8 weeks post-surgery
  Fat mass, fat-free mass, and percent body fat will be assessed using a whole-body scanner GE iDXA.
Body composition (by Magnetic Resonance Imaging (MRI)) | Change from baseline in body composition at 8 weeks post-surgery
  Visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT), and total adipose tissue (TAT) will be assessed by MRI scan (3T GE Discovery 750w).
Adipose tissue gene and protein expression | Changes from baseline in gene and protein expression at 8 weeks post-surgery
  Expression levels of genes and proteins involved in adipocyte expansion and function (ERα, PPARγ2, C/EBPα, aromatase, adiponectin, and LPL), extracellular matrix remodeling and fibrosis (COL6(a1, a2, a3), COL4a1, and TGFβ), and inflammation (IL-6 and TNFα) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Marlatt, PhD, MPH, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States